CLINICAL TRIAL: NCT07039565
Title: Efficacy of Combined Manual Diaphragm Release Technique and Neck Exercises in Adolescents With Forward Head Posture: a Randomized Controlled Trial
Brief Title: Efficacy of Combined Manual Diaphragm Release Technique and Neck Exercises in Adolescents With Forward Head Posture
Acronym: CVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Amal Youssef Wahba, Lecturer, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Treatment of forward head
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Forward Head Posture
Keywords: Manual diaphragm release technique; Postural assessment software (SAPO/PAS); adolescents; Forward head posture; Craniovertebral angle (CVA); Postural deviations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Manual diaphragm release technique and traditional neck exercises
  Interventions: Other: Stretching and strengthening exercises; Other: Diaphragm release technique
- Control group (Active Comparator): Traditional neck exercises
  Interventions: Other: Stretching and strengthening exercises

INTERVENTIONS:
Other: Stretching and strengthening exercises — Strengthening exercises were progressively performed for three sets, with 10 to 15 repetitions. The stretching part of the exercises was done with the purpose of increasing the flexibility of the pectoralis and the cervical neck extensors muscles (pectoralis stretch, chin tuck). Exercises have been approved to be effective on the lengthening of the pectoralis minor, activation of the lower trapezius/middle trapezius, serratus anterior, and improvement of the posture
Other: Diaphragm release technique — the patient will positioned in the supine position. The therapist stand at the head of the patient. The therapist make manual contact bilaterally under the costal cartilages of the lower ribs (7th to 10th ) with hypothenar regions of the hands and last three fingers. During the patient's inspiration, the therapist is gently pulling the points of hands contacts toward the head and slightly laterally, while elevating the ribs simultaneously
  Arms: Experimental group

SUMMARY:
* Due to the heavy use of smartphones among adolescents the cervical spine destabilizes and moves forward, so do the vital structures (nerves, arteries, veins) within the neck undergo torsion, stretch and compression including the autonomic nervous system nerves (which can cause dysfunction in heart rate, digestion, breathing among other symptoms).
* Forward head posture (FHP) puts more compressive strain on the cervical spine's tissues, especially the ligaments and facet joints. Because FHP weakens the respiratory muscles, it has a significant impact on respiratory function. Static balance may be negatively impacted by FHP.
* FHP is effectively treated by a proper and suitable physical therapy program.

DETAILED DESCRIPTION:
In the past few years, the number of smart phone users has progressively increased worldwide. With the growing use of smart phones, concerns have also increased about musculoskeletal problems associated with the prolonged use of smart phones.

Concerns have also increased about musculoskeletal problems associated with the prolonged use of smartphones. Recent investigations have shown that smartphone users tend to report pain in the neck, shoulder, and thumb, and the severity of the symptoms as the total time spent using the smartphone increases.

One of the most overspread postural abnormalities is forward head posture (FHP) and it is described as head projection anteriorly in relation to the trunk which appears mainly in sagittal plane. When using a smartphone, people usually flex their neck downwards to stare at the lowered object and maintain the head in a forward position for long periods of time, the maintenance of a head-forward posture decreases cervical lordosis of the lower cervical vertebrae and creates a posterior curve in the upper thoracic vertebrae to maintain balance; this is known as the forward head posture (FHP) that causes shortening of the extensors of the neck and producing chronic neck pain.

The weight supported by the spine dramatically increases when flexing the head forward at varying degrees. An adult head weighs 10-12 pounds in the neutral position. As the head tilts forward, the forces felt by the neck surge to 27 pounds at 15 degrees, 40 pounds at 30 degrees, 49 pounds at 45 degrees, and 60 pounds at 60 degrees. At 90 degrees, the model prediction was not reliable.

ELIGIBILITY:
Inclusion Criteria:

* Male students their age ranged from 17 to 18 years.
* Has Body Mass Index (BMI) = 5th percentile to less than the 85th percentile.

  _ has forward head posture
* Studying at any faculty at Pharos University in Alexandria.
* Cooperative and followed the instructions.

Exclusion Criteria:

* - Subjects were excluded from the study if the student had visual or hearing defects.
* Overweight, obese or cachexic students.
* Had any neurological disorders.
* Had musculoskeletal problems.
* Had any congenital abnormalities that might affect the study.

Ages: 17 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
craniovertebral angle (CVA) Forward head posture | 12 weeks
  The angle formed by a horizontal line crossing c7 and a line crossing c7 to the tragus of the ear is known as the CVA
Vertical head alignment (VHA) | 12 weeks
  Angle between right tragus, right acromion and vertical.

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa said Tolba, LecturerP, Study Chair — Pharos University in Alexandria; Amal Youssef Wahba, Lecturer, Principal Investigator — Pharos University in Alexandria
Locations (1):
- Pharos University in Alexandria, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Age, Degree of CVA, smart phone usage (hours/day)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 11/2025 - 5/2026
Access Criteria: Access through contacting E-mail: amal.youssef@pua.edu.eg
URL: https://amal.youssef@pua.edu.eg

REFERENCES:
- [Background] Lee KJ, Han HY, Cheon SH, Park SH, Yong MS. The effect of forward head posture on muscle activity during neck protraction and retraction. J Phys Ther Sci. 2015 Mar;27(3):977-9. doi: 10.1589/jpts.27.977. Epub 2015 Mar 31. PMID 25931773
- [Background] https://www.researchgate.net/publication/379140193_Forward_Head_Posture_and_Its_Effect_on_Muscle_Activation
- See also: Forward head posture (FHP), which is defined as a forward displacement of the head on the cervical spine, is a common postural disorder. It is suggested that this malalignment alters the loads on the spine, affects the length-tension relationship in musc — http://www.researchgate.net/publication/379140193_Forward_Head_Posture_and_Its_Effect_on_Muscle_Activation